CLINICAL TRIAL: NCT02532569
Title: A Multi-center, Open, phase4 Study to Assess the Long-term Immunogenicity and Safety of Fourth Administration of BR JEV and to Investigate on Vaccine Interchangeability in Children Aged 6 Years Who Received 3 Doses With ENCEVAC or JEV-GCC
Brief Title: Long-term Immunogenicity and Safety of Fourth Administration of Boryung Cell-Culture Japanese Encephalitis Vaccineinj
Acronym: BR-JELITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BR-KD-287-CT-401
Record Dates: First submitted 2015-08-21; First posted 2015-08-26 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Japanese encephalitis vaccine (Other): After reconstitution with 0.7 mL of the provided diluent, 0.5-mL dose,SC
  Interventions: Biological: Japanese encephalitis vaccine

INTERVENTIONS:
Biological: Japanese encephalitis vaccine — Dosage and administration: After reconstitution with 0.7 mL of the provided diluent, 0.5-mL dose is administered subcutaneously in the lateral aspect of the upper arm.
  Other Names: Boryung Cell-Culture Japanese Encephalitis Vaccine

SUMMARY:
A multi-center, open, phase 4 clinical trial to assess the long-term immunogenicity and safety of fourth administration of Boryung Cell-Culture Japanese Encephalitis Vaccine inj. and to conduct an exploratory investigation on vaccine interchangeability in Korean children aged 6 years who received primary 3 doses with ENCEVAC® or Japanese Encephalitis Vaccine-GCC® inj.

DETAILED DESCRIPTION:
This is a follow-up study of KD287-BR-CT-301 (ClinicalTrials.gov identifier: NCT01150942), a phase 3 study to investigate the efficacy and safety of a cell-culture Japanese encephalitis vaccine (ENCEVAC®) compared with that of a mouse brain-derived Japanese encephalitis vaccine (Japanese Encephalitis vaccine-GCC® inj). Subjects participated in KD287-BR-CT-301 study were to receive 3 doses of Japanese encephalitis vaccine (JEV) assigned by randomization from the age of 12 months and those subjects who completed the 3 doses of JEV are the target population in this study. The purpose of this study is to investigate the long-term immunogenicity and safety of the booster (fourth) dose of JEV, which will be given as Boryung Cell-Culture Japanese Encephalitis Vaccine inj, proven to be same with ENCEVAC® but manufactured by a different manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian (legally authorized representative) has given voluntary written consent to the subject's participation after being fully informed of the purpose, methods, risks, and benefits of the study.
* Male and female children who have completed the primary 3 doses of JEV in the KD287-BR-CT-301study.
* Male and female children reaching at least 6 years of age on the day of booster dosing of JEV.
* Male and female children who are identified to be healthy based on physical examination and medical history.

Exclusion Criteria:

* Children who have acute febrile illness with tympanic temperature of ≥38.0 ℃ on the day of booster dosing of JEV.
* Children who have moderate or severe acute disease (regardless of fever).
* Children who have history of encephalitis, encephalopathy, cerebromeningitis, or convulsion.
* Children who have received JEV (including live JEV) other than the investigational products administered in the KD287-BR-CT-301study.
* Children who have had fever (≥ 40 °C) or systemic allergy within 48 hours after vaccination.
* Children who have shown anaphylactic reaction to the investigational products administered in the KD287-BR-CT-301study or who are likely to be allergic to the ingredients of the investigational product.
* Children who have been diagnosed with immunodeficiency such as acquired immune deficiency or who have family history of immunodeficiency.
* Children who have received other vaccines within 28 days before booster dosing of JEV (vaccines to be administered according to the national vaccination program.
* Children who have received immunosuppressive thera-py within 28 days before booster dosing of JEV.
* There is a possibility that immune globulin preparations has not been excreted enough on the day of booster dosing of JEV if children have received such a product.
* Children who are currently participating or planning to participate in other clinical stud-ies during the study period.
* Other ineligible conditions judged at the discretion of principal investigators or subinvestigators.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To assess the seroconversion rates before and after the fourth dose of JEV | Day 28 (28 days after booster dose)]

SECONDARY OUTCOMES:
To assess the seropositive rates before and after the fourth dose of JEV | Day 28 (28 days after booster dose)]
To assess the geometric mean titer (GMT) before and after the fourth dose of JEV | Day 28 (28 days after booster dose)]
To assess the percentage of subjects who develop neutralizing antibody titers | Day 28 (28 days after booster dose)
To assess the percentage of subjects in their neutralizing anti-body titers | Day 28 (28 days after booster dose)

CONTACTS AND LOCATIONS:
Overall Officials: HJ Jung, MD, Study Director — Boryung Pharmaceutical Company
Locations (9):
- South Korea (9):
  - Wonju Sevrance Christian Hospital, Wŏnju, Gangwon-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
  - KyungHee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yun KW, Lee HJ, Park JY, Cho HK, Kim YJ, Kim KH, Kim NH, Hong YJ, Kim DH, Kim HM, Cha SH. Long-term immunogenicity of an initial booster dose of an inactivated, Vero cell culture-derived Japanese encephalitis vaccine (JE-VC) and the safety and immunogenicity of a second JE-VC booster dose in children previously vaccinated with an inactivated, mouse brain-derived Japanese encephalitis vaccine. Vaccine. 2018 Mar 7;36(11):1398-1404. doi: 10.1016/j.vaccine.2018.01.075. PMID 29429815